CLINICAL TRIAL: NCT03789383
Title: Risk Factors and Outcome of Biliary Complications Following Adult Living Donor Liver Transplantation in Al-Rajhy Liver Hospital in Upper Egypt.
Brief Title: Risk Factors and Outcome of Biliary Complications Following Adult Living Donor Liver Transplantation
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ali Hassan, Clinical teaching assistant in department of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: RFLTIUNE
Record Dates: First submitted 2018-12-25; First posted 2018-12-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplantation (LT) is a live-saving therapy for patients with complicated chronic liver diseases and acute liver failure .Even though many complications can occur after LT, biliary complications (BC) are both common and potentially severe .

a prospective study and retrospective part from hospital records.

Aim of the study:

1. Detect frequency, risk factors for development of biliary complications post living donor liver transplantation, types (stricture anastomotic or not, leak, biloma, stone, cholangitis etc.…).
2. Evaluate outcomes of different biliary complications

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 y with living donor liver transplantation in Al-Rajhy liver hospital , Assiut university,Egypt

Exclusion Criteria:

* pediatric liver transplantation
* cadaveric liver transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults more than 18 y with living donor liver transplantation in Al-Rajhy liver hospital, Assiut university, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of biliary complications | 1 year after liver transplantation
  Biliary complications include biliary leak or stricture (anastomotic or non anastomotic), the investigator will record nature of complication , its time of presentation and number of hospital re-admissions due to biliary complications.
Type of intervention done to each complication | 1 year after liver transplantation
  Intervention is either non surgical (ERCP or PTD) or surgical revision with detailed description of each intervention and if the intervention is successful or not (biliary stricture resolved by MRCP, improvement of liver functions and symptoms)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Alrajhy center for hepatobiliary disorders, Asyut
  - Al-Rajhy liver hospital, Asyut

IPD SHARING:
Plan to Share IPD: No